CLINICAL TRIAL: NCT03604939
Title: Improving Access to Control of Diseases for Women
Acronym: IMPACD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: GBH Cancer Memorial Hospital Udaipur, India (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DCA/SCR/2016/01
Record Dates: First submitted 2017-08-17; First posted 2018-07-30 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Cardio-vascular Disease; Stroke Cancer; Breast Cancer; Oral Cancer; Cervical Cancer
Keywords: cardio-vascular disease; stroke cancer; breast cancer; oral cancer; cervical cancer
MeSH Terms: conditions — Breast Neoplasms; Mouth Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: 35,000 households in 228 villages, among which women between 30 to 60 years residing in the villages of the block are eligible to participate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evaluation of social, cultural and behavioral factors — Evaluation of the social, cultural and behavioral factors that impact the uptake of the NCD prevention and control services among women, using the RARE methodology
Diagnostic Test: Evaluation of the feasibility and acceptability of delivery of early detections services — Evaluation of the feasibility and acceptability of delivery of the NCD early detections services by the trained community health workers at home settings

SUMMARY:
The aim of this study is to evaluate the feasibility and acceptability of the model of delivering CHW-driven home-based comprehensive NCD control services aimed to prevent premature deaths from cardio-vascular diseases, stroke and breast, cervix and oral cancers in the hard-to-reach women.

DETAILED DESCRIPTION:
Specific objectives of this study are the evaluation of:

1. The social, cultural and behavioral factors that impact the uptake of the NCD control services among rural women using the Rapid Assessment, Response and Evaluation (RARE) approach;
2. The feasibility and acceptability of the strategy to deliver the following NCD control services to the rural women at their homes by the trained CHWs:

   * Counselling of the tobacco habitués to give up the practice
   * Early detection of hypertension and diabetes to ensure prompt and regular treatment
   * Creating breast awareness and ensuring access to prompt diagnosis and treatment of the women with symptoms suggestive of breast cancer
   * Screening for cervical cancer by self-collected HPV test and ensuring prompt treatment of screen detected precancers and cancers
   * Screening of the habitual tobacco/alcohol users for oral cancer by OVE and ensuring prompt treatment of screen detected precancers and cancers

ELIGIBILITY:
Inclusion Criteria:

* Women between 30 to 60 years residing in the villages of the Gogunda block in the district of Udaipur in Rajasthan, India, will be eligible to participate.

Exclusion Criteria:

* Women suffering from debilitating illnesses, pregnant women and women refusing to participate will be excluded.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women between 30 to 60 years residing in the villages of the Gogunda block in the district of Udaipur in Rajasthan, India, will be eligible to participate.
Enrollment: 1200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Outcomes of the questionnaire survey 1/5 | 1 year
  proportion of the participants who know about the adverse effect of smoking, chewing tobacco and consuming alcohol on health in general and NCDs in particular
Outcomes of the questionnaire survey 2/5 | 1 year
  proportion of the participants who know about the common NCDs including cancers and their early symptoms
Outcomes of the questionnaire survey 3/5 | 1 year
  proportion of the participants with a diagnosis of hypertension who adhere to the treatment advised
Outcomes of the questionnaire survey 4/5 | 1 year
  proportion of the participants with a diagnosis of diabetes who adhere to the treatment advised
Outcomes of the questionnaire survey 5/5 | 1 year
  proportion of the participants with a diagnosis of cancer who adhere to the treatment advised
NCD Screening study 1/11 | 1 year
  screen positivity - proportion of the screened participants detected to have high blood pressure
NCD Screening study 2/11 | 1 year
  screen positivity - proportion of the screened participants detected to have high BMI
NCD Screening study 3/11 | 1 year
  screen positivity - proportion of the screened participants detected to have abnormal HPV detection test
NCD Screening study 4/11 | 1 year
  screen positivity - proportion of the screened participants detected to have abnormal oral examination test
NCD Screening study 5/11 | 1 year
  screen positivity - proportion of the screened participants detected to have abnormal visual examination test
NCD Screening study 6/11 | 1 year
  compliance to further assessment - proportion of screen positive participants undergoing further assessment at the primary health center or at the hospital
NCD Screening study 7/11 | 1 year
  positive predictive values of further assessment - proportion of participants with confirmed diagnosis of hypertension among those assessed for high BP
NCD Screening study 8/11 | 1 year
  positive predictive values of further assessment - proportion of participants with confirmed diabetes among those assessed for high sugar
NCD Screening study 9/11 | 1 year
  positive predictive values of further assessment - proportion of participants with confirmed cervical neoplasias on colposcopy and/or biopsy among those assessed for positive HPV test
NCD Screening study 10/11 | 1 year
  positive predictive values of further assessment - proportion of participants with confirmed oral premalignant and malignant lesions on examination and/or biopsy among those assessed for positive oral examination
NCD Screening study 11/11 | 1 year
  positive predictive values of further assessment - proportion of participants with confirmed visual premalignant and malignant lesions on examination and/or biopsy among those assessed for positive visual examination

SECONDARY OUTCOMES:
effect of different participant characteristics on the final diagnosis of hypertension and diabetes using multivariate analysis | 1 year
  effect of different participant characteristics on the final diagnosis of hypertension and diabetes using multivariate analysis

CONTACTS AND LOCATIONS:
Locations (1):
- GBH Cancer Memorial Hospital, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahajan M, Naik N, Jain K, Patira N, Prasad S, Mogri S, Muwonge R, Lucas E, Faruq F, Sankaranarayanan R, Iyer S, Basu P. Study of Knowledge, Attitudes, and Practices Toward Risk Factors and Early Detection of Noncommunicable Diseases Among Rural Women in India. J Glob Oncol. 2019 Apr;5:1-10. doi: 10.1200/JGO.18.00181. PMID 30998427
- [Background] Basu P, Mahajan M, Patira N, Prasad S, Mogri S, Muwonge R, Lucas E, Sankaranarayanan R, Iyer S, Naik N, Jain K. A pilot study to evaluate home-based screening for the common non-communicable diseases by a dedicated cadre of community health workers in a rural setting in India. BMC Public Health. 2019 Jan 3;19(1):14. doi: 10.1186/s12889-018-6350-4. PMID 30606132